CLINICAL TRIAL: NCT06911034
Title: Comparison of Ferric Carboxymaltose Versus Iron Sucrose for Treatment of Iron Deficiency Anemia in Pregnant Women
Brief Title: Ferric Carboxymaltose Versus Iron Sucrose for Treating Anemia in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CMH Multan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Kiran Saleem, Principal Investigator, CMH Multan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1319-2291
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Iron Deficiency Anemia (IDA); Pregnancy
Keywords: Iron deficiency anemia; Pregnancy; Ferric carboxymaltose; Iron sucrose
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose; Ferric Oxide, Saccharated; sucroferric oxyhydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carboxymaltose (Experimental): Intravenous infusion
  Interventions: Drug: Iron Carboxymaltose
- Sucrose (Active Comparator): Intravenous infusion
  Interventions: Drug: Iron Sucrose Injection

INTERVENTIONS:
Drug: Iron Carboxymaltose — In ferrous carboxymaltose treatment maximum dose per sitting was 1000 mg, diluted in 200 ml 0.9% normal saline and administered as an IV infusion over 30 min. Parenteral iron therapy was administered under doctor's supervision. The women were then followed up after 3 weeks of completion of therapy. On follow up, hemoglobin and serum ferritin were measured again.
  Other Names: Ferrous Carboxymaltose
  Arms: Carboxymaltose
Drug: Iron Sucrose Injection — Iron sucrose infusion was administered as 300 mg in 200 ml NS over 15-20 min twice weekly till dosage was completed, not exceeding 600 mg per week. Parenteral iron therapy was administered under doctor's supervision. The women were then followed up after 3 weeks of completion of therapy. On follow up, hemoglobin and serum ferritin were measured again.
  Other Names: sucroferric oxyhydroxide; Iron saccharate
  Arms: Sucrose

SUMMARY:
This clinical trial aimed to determine whether intravenous ferric carboxymaltose is more useful than iron sucrose for treating anemia in pregnant women.

The main question it aimed to answer was:

Is intravenous ferric carboxymaltose is more useful than iron sucrose for treating iron deficiency anemia in pregnant women.

Sixty pregnant women with iron deficiency anemia were enrolled to one of two intravenous treatments.

* Participants in ferrous carboxymaltose group received a maximum dose of 1000 mg per sitting diluted in 200 ml 0.9% normal saline and administered as an IV infusion over 30 min.
* Participants in iron sucrose group were administered an infusion of 300 mg in 200 ml NS over 15-20 min twice weekly till dosage was completed, not exceeding 600 mg per week.

DETAILED DESCRIPTION:
The study was conducted after the ethics review committee approval. A total of 60 pregnant women presenting to the department of Obstetrics and Gynecology and fulfilling the eligibility criteria were enrolled in the study after informed consent. Patient's characteristics including age, parity, area of residence, educational status, socioeconomic status and baseline Hb were recorded. All women were administered anthelminthic therapy with tablet mebendazole 100 mg twice daily for three days and given 5 mg Folic acid once daily. Patients were be randomly assigned to group A & B.

Patients in group A were treated with intravenous ferrous carboxymaltose and group B were given intravenous iron sucrose complex. Parenteral iron therapy was administered under doctor's supervision. The women were then followed up after 3 weeks of completion of therapy. On follow up, hemoglobin and serum ferritin were measured again.

ELIGIBILITY:
Inclusion Criteria:

* 28-34 weeks of gestation
* Iron deficiency anemia (IDA): IDA will be labelled if Hemoglobin is <10 gm% and serum Ferritin < 30 ng/ml.

Exclusion Criteria:

* Hepatitis (serum transaminases more than 1.5 times the upper limit of normal) and HIV infection
* serum creatinine level of more than 2.0 mg/dL
* history of allergic reaction to intravenous iron infusion

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | After three weeks of completing parenteral iron therapy
  Rise in hemoglobin (g/dl) will be calculated by subtracting post treatment hemoglobin from pre-treatment hemoglobin

SECONDARY OUTCOMES:
Ferritin levels | Three weeks after completion of parenteral iron therapy
  Post treatment ferritin levels will be done

CONTACTS AND LOCATIONS:
Overall Officials: Nidda Ya Consultant, FCPS, Study Chair — CMH Multan Institute of Medical Sciences
Locations (1):
- Cmh Multan Institute of Medical Sciences, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Sharing IPD can compromise patient privacy, even if identifying details are removed. Sensitive medical information could potentially be re-identified, violating ethical guidelines.

REFERENCES:
- [Background] Bharadwaj MK, Patrikar S, Singh Y. Comparative analysis of injection ferric carboxymaltose vs iron sucrose for treatment of iron-deficiency anemia in pregnancy: systematic review and meta-analysis. J South Asian Fed Obstet Gynaecol. 2023;15(5):629-36.
- [Background] Comparison of ferric carboxymaltose and iron sucrose for treatment of iron deficiency anemia in pregnancy at tertiary care centre, Western India. Int J Reprod Contracept Obstet Gynecol. 2023;12(6):1844-8.
- [Background] Jose A, Mahey R, Sharma JB, Bhatla N, Saxena R, Kalaivani M, Kriplani A. Comparison of ferric Carboxymaltose and iron sucrose complex for treatment of iron deficiency anemia in pregnancy- randomised controlled trial. BMC Pregnancy Childbirth. 2019 Feb 4;19(1):54. doi: 10.1186/s12884-019-2200-3. PMID 30717690